CLINICAL TRIAL: NCT01634139
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate Efficacy and Safety of Tiotropium Inhalation Solution (2.5 mcg and 5 mcg) Delivered Via Respimat® Inhaler Once Daily in the Evening Over 48 Weeks in Children (6 to 11 Years Old) With Moderate Persistent Asthma
Brief Title: Efficacy and Safety of 2 Doses of Tiotropium Respimat® Compared to Placebo in Children With Moderate Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.445; 2011-001758-26 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (3):
- Tiotropium high dose QD (Experimental)
  Interventions: Drug: Tiotropium high dose QD
- Tiotropium low dose QD (Experimental)
  Interventions: Drug: Tiotropium low dose QD
- Placebo QD (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium low dose QD — 2 actuations once daily in the evening
  Arms: Tiotropium low dose QD
Drug: Tiotropium high dose QD — 2 actuations once daily in the evening
  Arms: Tiotropium high dose QD
Drug: Placebo — 2 actuations once daily in the evening
  Arms: Placebo QD

SUMMARY:
The overall purpose of the trial is to evaluate efficacy and safety of tiotropium inhalation solution delivered via Respimat® inhaler (2.5 mcg and 5 mcg once daily in the evening) over 48 weeks, compared to placebo, in children (6 to 11 years old) with moderate persistent asthma.

ELIGIBILITY:
Inclusion criteria:

Inclusion criteria are:

1. All patients' parent(s) (or legal guardian) must sign and date an informed consent prior to participation in the trial. In addition, an informed assent suitable for this age group has to be obtained from patients. A separate informed consent/assent is required for pharmacogenomic sampling.
2. Male or female patients between 6 and 11 years of age.
3. All patients must have at least a 6-month history of asthma.
4. All patients must have been on maintenance treatment with an inhaled corticosteroid at a stable medium dose, either as mono treatment or in combination with another controller medication, for at least 4 weeks before Visit 1. While the LTRA is permitted throughout the trial, the LABA has to be stopped at least 24 hours prior to Visit 1, as no LABAs are permitted during screening and treatment period of this trial.
5. All patients must be symptomatic (partly controlled) at Visit 1 and prior to randomisation at Visit 2 as defined by an Asthma Control Questionnaire (ACQ-IA) mean score >= 1.5.
6. All patients must have a pre-bronchodilator forced expiratory volume in one second (FEV1) >= 60% and =< 90% of predicted normal at Visit 1.
7. Variation of absolute FEV1 values of Visit 1 (pre-bronchodilator, considered as 100%) as compared to Visit 2 (pre-dose) must be within ± 30%.
8. All patients must confirm the diagnosis of asthma by bronchodilator reversibility at Visit 1, resulting in an increase in FEV1 of >= 12%, 15 to 30 minutes after 200 mcg salbutamol/albuterol.
9. Patients must be able to use the Respimat inhaler correctly.
10. Patients must be able to perform all trial related procedures including technically acceptable pulmonary function tests and use of electronic diary/peak flow meter (diary compliance of at least 80% is required).

Exclusion criteria:

Exclusion criteria are:

1. Patients with a significant disease other than asthma.
2. Patients with a clinically relevant abnormal haematology or blood chemistry at screening.
3. Patients with a history of congenital or acquired heart disease, or patients who have been hospitalized for cardiac syncope or failure during the past year.
4. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
5. Patients with a malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years.
6. Patients with known active tuberculosis.
7. Patients who have undergone thoracotomy with pulmonary resection.
8. Patients who are currently in a pulmonary rehabilitation program or have completed a pulmonary rehabilitation program in the six weeks prior to Visit 1.
9. Patients with known hypersensitivity to anticholinergic drugs, BAC, EDTA or any other components of the inhalation solution used with the Respimat inhaler.
10. Pregnant or nursing female patients, including postmenarchal girl with a positive urine pregnancy test at Visit 1.
11. Postmenarchal girl of child-bearing potential not using a highly effective method of birth control.
12. Patients who have been treated with anti-IgE treatment within the last six months prior to Visit 1 and/or during the screening period.
13. Patients who have been treated with systemic corticosteroids within four weeks prior to Visit 1.
14. Patients who have been treated with systemic beta-adrenergics within four weeks prior to Visit 1.
15. Patients who have been treated with oral beta-blocker medication within four weeks prior to Visit 1 and/or during the screening period.
16. Patients who have been treated with inhaled long-acting anticholinergics or systemic anticholinergic treatment within four weeks prior to Visit 1 and/or during the screening period or who have been treated with inhaled short-acting anticholinergics within two weeks prior to Visit 1.
17. Patients who have been treated with long-acting theophylline preparations within four weeks prior to Visit 1 and/or during the screening period or who have been treated with short-acting theophylline preparations within two weeks prior to Visit 1.
18. Patients who have been treated with non-approved and according to international guidelines not recommended experimental drugs for routine asthma therapy within four weeks prior to Visit 1 and/or during the screening period.
19. Patients who have taken an investigational drug within six half lives according to the investigator's information, or four weeks (whichever is greater) prior to Visit 1 and/or during the screening period.
20. Patients who have previously been randomised in this trial or are currently participating in another trial.
21. Patients with any acute asthma exacerbation or respiratory tract infection in the four weeks prior to Visit 1 and /or in four weeks prior to Visit 2. In case of an asthma deterioration occurring in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2, the visit must be postponed.
22. Patients requiring six or more puffs of rescue medication per day on more than two consecutive days in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2. In case of an asthma deterioration occurring in the four weeks prior to Visit 1 and/or in the four weeks prior to Visit 2, the visit must be postponed.
23. Patients who are unable to comply with medication restrictions prior to Visit 1 and or Visit 2.
24. Patients with a known narrow-angle glaucoma, or any other disease where anticholinergic treatment is contraindicated.
25. Patients with moderate to severe renal impairment, as defined by a creatinine clearance <50 mL/min/1.73 m2 BSA, as tiotropium is a predominantly renally excreted drug.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 403 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (79):
- United States (6):
  - 205.445.01002 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 205.445.01001 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.445.01010 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 205.445.01006 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 205.445.01012 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 205.445.01004 Boehringer Ingelheim Investigational Site, El Paso, Texas
- Bulgaria (5):
  - 205.445.35901 Boehringer Ingelheim Investigational Site, Sofia
  - 205.445.35902 Boehringer Ingelheim Investigational Site, Sofia
  - 205.445.35903 Boehringer Ingelheim Investigational Site, Sofia
  - 205.445.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 205.445.35905 Boehringer Ingelheim Investigational Site, Sofia
- Canada (2):
  - 205.445.02003 Boehringer Ingelheim Investigational Site, London, Ontario
  - 205.445.02001 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
- Germany (7):
  - 205.445.49012 Boehringer Ingelheim Investigational Site, Berlin
  - 205.445.49015 Boehringer Ingelheim Investigational Site, Berlin
  - 205.445.49001 Boehringer Ingelheim Investigational Site, Bochum
  - 205.445.49007 Boehringer Ingelheim Investigational Site, Dresden
  - 205.445.49004 Boehringer Ingelheim Investigational Site, Ettenheim
  - 205.445.49009 Boehringer Ingelheim Investigational Site, Koblenz
  - 205.445.49014 Boehringer Ingelheim Investigational Site, Marburg
- Guatemala (5):
  - 205.445.50201 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.445.50202 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.445.50203 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.445.50204 Boehringer Ingelheim Investigational Site, Guatemala City
  - 205.445.50205 Boehringer Ingelheim Investigational Site, Guatemala City
- Hungary (3):
  - 205.445.36003 Boehringer Ingelheim Investigational Site, Ajka
  - 205.445.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 205.445.36002 Boehringer Ingelheim Investigational Site, Dombóvár
- Latvia (8):
  - 205.445.37104 Boehringer Ingelheim Investigational Site, Ādaži
  - 205.445.37101 Boehringer Ingelheim Investigational Site, Baldone
  - 205.445.37106 Boehringer Ingelheim Investigational Site, Balvi
  - 205.445.37108 Boehringer Ingelheim Investigational Site, Daugavpils
  - 205.445.37102 Boehringer Ingelheim Investigational Site, Ogre
  - 205.445.37107 Boehringer Ingelheim Investigational Site, Rēzekne
  - 205.445.37103 Boehringer Ingelheim Investigational Site, Riga
  - 205.445.37105 Boehringer Ingelheim Investigational Site, Riga
- Lithuania (3):
  - 205.445.37002 Boehringer Ingelheim Investigational Site, Šiauliai
  - 205.445.37005 Boehringer Ingelheim Investigational Site, Utena
  - 205.445.37003 Boehringer Ingelheim Investigational Site, Vilnius
- 205.445.47002 Boehringer Ingelheim Investigational Site, Oslo, Norway
- Portugal (7):
  - 205.445.35108 Boehringer Ingelheim Investigational Site, Amadora
  - 205.445.35106 Boehringer Ingelheim Investigational Site, Aveiro
  - 205.445.35101 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.445.35102 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.445.35107 Boehringer Ingelheim Investigational Site, Lisbon
  - 205.445.35103 Boehringer Ingelheim Investigational Site, Porto
  - 205.445.35105 Boehringer Ingelheim Investigational Site, Porto
- Romania (3):
  - 205.445.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.445.40004 Boehringer Ingelheim Investigational Site, Bucharest
  - 205.445.40003 Boehringer Ingelheim Investigational Site, Cluj-Napoca
- Russia (9):
  - 205.445.70002 Boehringer Ingelheim Investigational Site, Moscow
  - 205.445.70005 Boehringer Ingelheim Investigational Site, Moscow
  - 205.445.70008 Boehringer Ingelheim Investigational Site, Moscow
  - 205.445.70011 Boehringer Ingelheim Investigational Site, Moscow
  - 205.445.70001 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.445.70003 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.445.70004 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.445.70009 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 205.445.70010 Boehringer Ingelheim Investigational Site, Yaroslavl
- South Korea (5):
  - 205.445.82003 Boehringer Ingelheim Investigational Site, Guri-si
  - 205.445.82002 Boehringer Ingelheim Investigational Site, Incheon
  - 205.445.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 205.445.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 205.445.82006 Boehringer Ingelheim Investigational Site, Sungnam
- 205.445.46001 Boehringer Ingelheim Investigational Site, Stockholm, Sweden
- Ukraine (13):
  - 205.445.38017 Boehringer Ingelheim Investigational Site, Chernivtsi
  - 205.445.38003 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 205.445.38005 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.445.38011 Boehringer Ingelheim Investigational Site, Donetsk
  - 205.445.38008 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.445.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 205.445.38012 Boehringer Ingelheim Investigational Site, Kryvyi Rih
  - 205.445.38001 Boehringer Ingelheim Investigational Site, Lviv
  - 205.445.38009 Boehringer Ingelheim Investigational Site, Lviv
  - 205.445.38016 Boehringer Ingelheim Investigational Site, Odesa
  - 205.445.38006 Boehringer Ingelheim Investigational Site, Vinnytsia
  - 205.445.38010 Boehringer Ingelheim Investigational Site, Zaporizhya
  - 205.445.38002 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- 205.445.44001 Boehringer Ingelheim Investigational Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Respimat: Inhalation of placebo solution (2 puffs) once daily for 48 weeks delivered by the Respimat inhaler, as add on therapy on top of usual care.
- Tio R2.5: Inhalation of 2.5mcg tiotropium (Tio R2.5) solution (2 puffs of 1.25mcg) once daily for 48 weeks delivered by the Respimat inhaler, as add on therapy on top of usual care.
- Tio R5: Inhalation of 5mcg tiotropium (Tio R5) solution (2 puffs of 2.5mcg) once daily for 48 weeks delivered by the Respimat inhaler, as add on therapy on top of usual care.
Period: Overall Study
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Started | 132 | 136 | 135
Completed | 122 | 130 | 130
Not Completed | 10 | 6 | 5
Not completed — Non compliant with protocol | 1 | 0 | 0
Not completed — Consent withdrawn not due to AE | 4 | 3 | 2
Not completed — Other | 4 | 0 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Not treated | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This patient set included all randomised patients who were dispensed study medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5 | Total
Number analyzed (Participants) | 131 | 135 | 135 | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.0 (1.6) | 9.0 (1.6) | 8.9 (1.7) | 8.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 38 | 53 | 137
  Male | 85 | 97 | 82 | 264

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Peak (0-3h) Change From Baseline
Description: Change from baseline in peak forced expiratory volume (FEV) in 1 second within the first 3 hours (h) post dosing (FEV1 peak(0-3h)) measured at week 24.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Time Frame: Baseline and 24 Weeks.
Population: Full Analysis Set (FAS) was equal to treated set which included all randomised patients who received at least 1 documented dose of study medication. Missing data at a visit was imputed by available data from the patient at that visit. Completely missing data were handled by the statistical model.
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 126 | 131 | 134
Litres (L) | 0.225 (0.027) | 0.395 (0.026) | 0.389 (0.026)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Stepwise testing of the null hypothesis was used to test the efficacy of Tio R5 and then Tio R2.5, each over placebo. The analysis was performed in a stepwise manner, firstly for this endpoint, then Trough FEV1. Each step was only considered confirmatory if all previous steps were successful; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.170, 95% CI 2-sided [0.108 to 0.231], Standard Error of Mean 0.031 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.164, 95% CI 2-sided [0.103 to 0.255], Standard Error of Mean 0.031 — Difference calculated as Tio R5 minus placebo

2. Secondary Outcome: Trough FEV1 Change From Baseline
Description: Change from Baseline in Trough (pre-dose) Forced Expiratory Volume (FEV) in 1 second (FEV1) measured at week 24 and 48.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres (L)
  Week 24 (N=126, 131, 134) | 0.156 (0.031) | 0.272 (0.030) | 0.274 (0.030)
  Week 48 (N=124, 130, 130) | 0.266 (0.032) | 0.337 (0.030) | 0.365 (0.031)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.116, 95% CI 2-sided [0.046 to 0.186], Standard Error of Mean 0.036 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.118, 95% CI 2-sided [0.048 to 0.188], Standard Error of Mean 0.036 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.0477, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.071, 95% CI 2-sided [0.001 to 0.142], Standard Error of Mean 0.036 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.0059, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.099, 95% CI 2-sided [0.029 to 0.170], Standard Error of Mean 0.036 — Difference calculated as Tio R5 minus placebo

3. Secondary Outcome: FEV1 Peak (0-3h) at Week 48 Change From Baseline
Description: Change from baseline in peak forced expiratory volume (FEV) in 1 second within the first 3 hours (h) post dosing (FEV1 peak(0-3h)) measured at week 48.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Time Frame: Baseline and Week 48.
Population: FAS. Missing data at a visit was imputed by available data from the patient at that visit. Completely missing data were handled by the statistical model.
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 124 | 130 | 130
Litres (L) | 0.351 (0.027) | 0.474 (0.026) | 0.477 (0.026)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.124, 95% CI 2-sided [0.062 to 0.185], Standard Error of Mean 0.031 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.127, 95% CI 2-sided [0.065 to 0.188], Standard Error of Mean 0.031 — Difference calculated as Tio R5 minus placebo

4. Secondary Outcome: FEV1 AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 hours for FEV1 (FEV1 AUC (0-3h)) after 24 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at week 24
Population: FAS, missing data at a visit was imputed by the available data from the patient at that visit. Completely missing data were handled by the statistical model.
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 126 | 131 | 134
Litres (L) | 0.152 (0.026) | 0.306 (0.025) | 0.309 (0.025)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.154, 95% CI 2-sided [0.095 to 0.212], Standard Error of Mean 0.030 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.157, 95% CI 2-sided [0.098 to 0.215], Standard Error of Mean 0.030 — Difference calculated as Tio R5 minus placebo

5. Secondary Outcome: FEV1 Change From Baseline at Each Individual Timepoint
Description: FEV1 change from baseline to week 24 at each individual timepoint.
  The measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 24 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres (L)
  10 minutes pre-dose (Week 24) (N=126, 131, 134) | 0.156 (0.031) | 0.272 (0.030) | 0.274 (0.030)
  30 minutes post-dose (Week 24) (N=126, 131, 134) | 0.156 (0.027) | 0.295 (0.026) | 0.307 (0.027)
  1 hour post-dose (Week 24) (N=126, 131, 134) | 0.165 (0.028) | 0.313 (0.027) | 0.312 (0.027)
  2 hours post-dose (Week 24) (N=126, 131, 134) | 0.144 (0.028) | 0.307 (0.027) | 0.312 (0.027)
  3 hours post-dose (Week 24) (N=126, 131, 134) | 0.147 (0.027) | 0.325 (0.026) | 0.322 (0.026)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; 10 minutes pre-dose (Week 24); Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.116, 95% CI 2-sided [0.046 to 0.186], Standard Error of Mean 0.036 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; 10 minutes pre-dose (Week 24); Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.118, 95% CI 2-sided [0.048 to 0.188], Standard Error of Mean 0.036 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; 30 minutes post-dose (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.139, 95% CI 2-sided [0.076 to 0.201], Standard Error of Mean 0.032 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; 30 minutes post-dose (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.151, 95% CI 2-sided [0.088 to 0.213], Standard Error of Mean 0.032 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 5: Comparison: Placebo Respimat vs Tio R2.5; 1 hour post-dose (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.148, 95% CI 2-sided [0.084 to 0.211], Standard Error of Mean 0.032 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 6: Comparison: Placebo Respimat vs Tio R5; 1 hour post-dose (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.147, 95% CI 2-sided [0.084 to 0.210], Standard Error of Mean 0.032 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 7: Comparison: Placebo Respimat vs Tio R2.5; 2 hours post-dose (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.163, 95% CI 2-sided [0.101 to 0.226], Standard Error of Mean 0.032 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 8: Comparison: Placebo Respimat vs Tio R5; 2 hours post-dose (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.168, 95% CI [0.106 to 0.231], Standard Error of Mean 0.032 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 9: Comparison: Placebo Respimat vs Tio R2.5; 3 hours post-dose (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.178, 95% CI 2-sided [0.116 to 0.240], Standard Error of Mean 0.032 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 10: Comparison: Placebo Respimat vs Tio R5; 3 hours post-dose (Week 24); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.176, 95% CI 2-sided [0.114 to 0.238], Standard Error of Mean 0.032 — Difference calculated as Tio R5 minus placebo

6. Secondary Outcome: FVC Peak(0-3h) Change From Baseline
Description: Change from baseline in Maximum forced vital capacity (FVC) measured within the first 3 hours after administration of trial medication (FVC peak(0-3h)) after 24 and 48 Weeks of treatment.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres (L)
  Week 24 (N=124, 130, 134) | 0.215 (0.033) | 0.325 (0.032) | 0.307 (0.032)
  Week 48 (N=124, 130, 130) | 0.361 (0.033) | 0.430 (0.032) | 0.413 (0.032)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0036, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.110, 95% CI 2-sided [0.036 to 0.184], Standard Error of Mean 0.038 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0152, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.091, 95% CI 2-sided [0.018 to 0.165], Standard Error of Mean 0.037 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.0687, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.069, 95% CI 2-sided [-0.005 to 0.143], Standard Error of Mean 0.038 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.1666, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.052, 95% CI 2-sided [-0.022 to 0.126], Standard Error of Mean 0.038 — Difference calculated as Tio R5 minus placebo

7. Secondary Outcome: Trough FVC Change From Baseline
Description: Change from baseline in Trough (pre-dose) FVC measured at week 24 and 48.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres (L)
  Week 24 (N=126, 131, 134) | 0.154 (0.035) | 0.246 (0.034) | 0.206 (0.034)
  Week 48 (N=124, 130, 130) | 0.280 (0.035) | 0.341 (0.034) | 0.333 (0.034)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0228, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.092, 95% CI 2-sided [0.013 to 0.171], Standard Error of Mean 0.040 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.1980, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.052, 95% CI 2-sided [-0.027 to 0.131], Standard Error of Mean 0.040 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.1256, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.062, 95% CI 2-sided [-0.017 to 0.141], Standard Error of Mean 0.040 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.1880, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.053, 95% CI 2-sided [-0.026 to 0.133], Standard Error of Mean 0.040 — Difference calculated as Tio R5 minus placebo

8. Secondary Outcome: FVC AUC (0-3h) Change From Baseline
Description: Change from baseline of area under the curve (AUC) from 0 to 3 hours for FVC (Forced vital capacity) (FVC AUC (0-3h)) after 24 weeks of treatment. The AUC was calculated by using the trapezoidal rule divided by the observation time (3h).
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants with available data at the timepoint of interest.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at 24 weeks
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 126 | 131 | 134
Litres (L) | 0.130 (0.030) | 0.235 (0.029) | 0.207 (0.029)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.105, 95% CI 2-sided [0.037 to 0.172], Standard Error of Mean 0.034 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0255, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.076, 95% CI 2-sided [0.009 to 0.143], Standard Error of Mean 0.034 — Difference calculated as Tio R5 minus placebo

9. Secondary Outcome: FVC Change From Baseline at Each Individual Timepoint
Description: FVC change from baseline to week 24 at each individual timepoint.
  The measured values presented are actually adjusted means
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and 10 mins before drug administration and 30 mins, 1 hour (h), 2h, 3h after drug administration at Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres (L)
  10 minutes pre-dose (Week 24) (N=124, 131, 134) | 0.154 (0.035) | 0.246 (0.034) | 0.206 (0.034)
  30 minutes post-dose (Week 24) (N=124, 131, 134) | 0.144 (0.032) | 0.222 (0.031) | 0.211 (0.031)
  1 hour post-dose (Week 24) (N=124, 131, 134) | 0.142 (0.032) | 0.252 (0.031) | 0.202 (0.031)
  2 hours post-dose (Week 24) (N=124, 131, 134) | 0.117 (0.033) | 0.230 (0.031) | 0.210 (0.032)
  3 hours post-dose (Week 24) (N=124, 131, 134) | 0.118 (0.033) | 0.233 (0.032) | 0.210 (0.032)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; 10 minutes pre-dose (Week 24); Test type: Superiority or Other; p = 0.0228, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.092, 95% CI 2-sided [0.013 to 0.171], Standard Error of Mean 0.040 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; 10 minutes pre-dose.(Week 24); Test type: Superiority or Other; p = 0.1980, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.052, 95% CI 2-sided [-0.027 to 0.131], Standard Error of Mean 0.040 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; 30 minutes post-dose (Week 24); Test type: Superiority or Other; p = 0.0344, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.078, 95% CI 2-sided [0.006 to 0.150], Standard Error of Mean 0.037 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; 30 minutes post-dose (Week 24); Test type: Superiority or Other; p = 0.0696, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.067, 95% CI 2-sided [-0.005 to 0.139], Standard Error of Mean 0.037 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 5: Comparison: Placebo Respimat vs Tio R2.5; 1 hour post-dose (week 24); Test type: Superiority or Other; p = 0.0032, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.109, 95% CI 2-sided [0.037 to 0.182], Standard Error of Mean 0.037 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 6: Comparison: Placebo Respimat vs Tio R5; 1 hour post-dose (week 24); Test type: Superiority or Other; p = 0.1044, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.060, 95% CI 2-sided [-0.012 to 0.132], Standard Error of Mean 0.037 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 7: Comparison: Placebo Respimat vs Tio R2.5; 2 hours post-dose (week 24); Test type: Superiority or Other; p = 0.0027, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.113, 95% CI 2-sided [0.039 to 0.186], Standard Error of Mean 0.037 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 8: Comparison: Placebo Respimat vs Tio R5; 2 hours post-dose (week 24); Test type: Superiority or Other; p = 0.0130, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.093, 95% CI 2-sided [0.020 to 0.166], Standard Error of Mean 0.037 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 9: Comparison: Placebo Respimat vs Tio R2.5; 3 hours post-dose (week 24); Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.115, 95% CI 2-sided [0.041 to 0.190], Standard Error of Mean 0.038 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 10: Comparison: Placebo Respimat vs Tio R5; 3 hours post-dose (Week 24); Test type: Superiority or Other; p = 0.0156, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.092, 95% CI 2-sided [0.017 to 0.166], Standard Error of Mean 0.038 — Difference calculated as Tio R5 minus placebo

10. Secondary Outcome: Use of PRN (Pro re Nata) Rescue Medication Per Day
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used per day (24 hour period) based on the weekly mean at weeks 24 and 48.
  The measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Number of puffs of rescue medication
  Week 24 (N=122, 130, 133) | -0.437 (0.079) | -0.603 (0.077) | 0.646 (0.077)
  Week 48 (N=120, 123, 127) | -0.484 (0.079) | 0.638 (0.078) | 0.685 (0.078)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.1349, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.165, 95% CI 2-sided [-0.382 to 0.051], Standard Error of Mean 0.110 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0588, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.209, 95% CI 2-sided [-0.425 to 0.008], Standard Error of Mean 0.110 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.1675, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.154, 95% CI 2-sided [-0.372 to 0.065], Standard Error of Mean 0.111 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.0709, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.201, 95% CI 2-sided [-0.419 to 0.017], Standard Error of Mean 0.111 — Difference calculated as Tio R5 minus placebo

11. Secondary Outcome: Use of PRN Rescue Medication During Daytime
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during daytime based on the weekly mean at weeks 24 and 48.
  Measured values presented are actually adjusted means
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Number of puffs of rescue medication
  Week 24 (N=121, 130, 133) | -0.234 (0.055) | -0.350 (0.053) | -0.375 (0.053)
  Week 48 (N=119, 123, 125) | -0.247 (0.055) | -0.372 (0.053) | -0.378 (0.053)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0749, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.116, 95% CI 2-sided [-0.245 to 0.012], Standard Error of Mean 0.065 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0305, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.141, 95% CI 2-sided [-0.269 to -0.013], Standard Error of Mean 0.065 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.0581, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.125, 95% CI 2-sided [-0.255 to 0.004], Standard Error of Mean 0.066 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.0464, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.131, 95% CI 2-sided [-0.260 to -0.002], Standard Error of Mean 0.066 — Difference calculated as Tio R5 minus placebo

12. Secondary Outcome: Use of PRN Rescue Medication During Nighttime
Description: Change from baseline in the number of puffs of rescue medication (salbutamol/albuterol) used during nighttime based on the weekly mean at weeks 24 and 48.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Number of puffs of rescue medication
  Week 24 (N=122, 130, 130) | -0.178 (0.051) | -0.274 (0.050) | -0.304 (0.050)
  Week 48 (N=119, 122, 125) | -0.198 (0.052) | -0.298 (0.050) | -0.301 (0.050)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.1182, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.096, 95% CI 2-sided [-0.217 to 0.025], Standard Error of Mean 0.062 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0404, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.126, 95% CI 2-sided [-0.246 to -0.006], Standard Error of Mean 0.061 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.1105, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.099, 95% CI 2-sided [-0.221 to 0.023], Standard Error of Mean 0.062 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.0983, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.103, 95% CI 2-sided [-0.224 to 0.019], Standard Error of Mean 0.062 — Difference calculated as Tio R5 minus placebo

13. Secondary Outcome: Peak Expiratory Flow (PEF) a.m. Change From Baseline
Description: Change from baseline in the morning (a.m.) peak expiratory flow based on the weekly mean at weeks 24 and 48.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres per min (L/min)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres per min (L/min)
  Week 24 (N=122, 130, 130) | 14.153 (4.556) | 22.660 (4.406) | 21.646 (4.434)
  Week 48 (N=119, 122, 125) | 20.824 (4.581) | 26.362 (4.440) | 29.598 (4.466)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.1146, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 8.507, 95% CI 2-sided [-2.063 to 19.077], Standard Error of Mean 5.387 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.1628, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 7.493, 95% CI 2-sided [-3.034 to 18.020], Standard Error of Mean 5.365 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.3085, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 5.538, 95% CI 2-sided [-5.127 to 16.203], Standard Error of Mean 5.435 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.1053, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 8.774, 95% CI 2-sided [-1.847 to 19.394], Standard Error of Mean 5.413 — Difference calculated as Tio R5 minus placebo

14. Secondary Outcome: PEF p.m. Change From Baseline
Description: Change from baseline in the evening (p.m.) peak expiratory flow based on the weekly mean at weeks 24 and 48.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres per min (L/min)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres per min (L/min)
  Week 24 (N= 121, 130, 133) | 3.179 (4.597) | 15.539 (4.444) | 17.325 (4.464)
  Week 48 (N=119, 123, 125) | 17.100 (4.622) | 15.219 (4.475) | 21.276 (4.504)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0236, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 12.360, 95% CI 2-sided [1.663 to 23.056], Standard Error of Mean 5.451 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0093, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 14.146, 95% CI 2-sided [3.497 to 24.794], Standard Error of Mean 5.427 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.7322, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -1.882, 95% CI 2-sided [-12.667 to 8.904], Standard Error of Mean 5.497 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.4463, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 4.176, 95% CI 2-sided [-6.578 to 14.929], Standard Error of Mean 5.481 — Difference calculated as Tio R5 minus placebo

15. Secondary Outcome: PEF Variability Change From Baseline
Description: Change from baseline in the peak expiratory flow variability based on the weekly mean at week 24 and 48.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Percentage of PEF
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Percentage of PEF
  Week 24 (N=121, 129, 128) | -1.204 (0.826) | -0.942 (0.798) | -1.038 (0.803)
  Week 48 (N=117, 120, 121) | -0.320 (0.835) | -0.048 (0.814) | -0.899 (0.818)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.8008, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.262, 95% CI 2-sided [-1.775 to 2.299], Standard Error of Mean 1.039 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.8731, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.166, 95% CI 2-sided [-1.875 to 2.208], Standard Error of Mean 1.041 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.7975, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.272, 95% CI 2-sided [-1.803 to 2.346], Standard Error of Mean 1.058 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.5845, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.579, 95% CI 2-sided [-2.656 to 1.498], Standard Error of Mean 1.059 — Difference calculated as Tio R5 minus placebo

16. Secondary Outcome: FEV1 a.m Change From Baseline
Description: Change from baseline in morning (a.m.) FEV1 based on the weekly mean at week 24 and 48.
  The measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres
  Week 24 (N=122, 130, 130) | 0.191 (0.041) | 0.209 (0.039) | 0.126 (0.039)
  Week 48 (N=119, 122, 125) | 0.236 (0.041) | 0.259 (0.040) | 0.221 (0.040)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.6932, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.019, 95% CI 2-sided [-0.075 to 0.113], Standard Error of Mean 0.048 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.1741, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.065, 95% CI 2-sided [-0.158 to 0.029], Standard Error of Mean 0.048 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.6250, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.024, 95% CI 2-sided [-0.071 to 0.118], Standard Error of Mean 0.048 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.7597, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.015, 95% CI 2-sided [-0.109 to 0.080], Standard Error of Mean 0.048 — Difference calculated as Tio R5 minus placebo

17. Secondary Outcome: FEV1 p.m. Change From Baseline
Description: Change from baseline in evening (p.m.) FEV1 based on the weekly mean at week 24 and 48.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Litres (L)
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Litres (L)
  Week 24 (N=121, 129, 128) | 0.167 (0.042) | 0.142 (0.041) | 0.092 (0.041)
  Week 48 (N=119, 123, 125) | 0.202 (0.042) | 0.208 (0.041) | 0.159 (0.041)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.6166, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.025, 95% CI 2-sided [-0.122 to 0.073], Standard Error of Mean 0.050 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.1267, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.076, 95% CI 2-sided [-0.173 to 0.021], Standard Error of Mean 0.049 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.9000, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.006, 95% CI 2-sided [-0.092 to 0.105], Standard Error of Mean 0.050 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.3897, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.043, 95% CI 2-sided [-0.141 to 0.055], Standard Error of Mean 0.050 — Difference calculated as Tio R5 minus placebo

18. Secondary Outcome: ACQ-IA Total Score
Description: Interviewer Administered Asthma Control Questionnaire (ACQ-IA) total score after 24 and 48 weeks of treatment.
  The ACQ-IA is a scale containing 7 questions. Each question has a 7 point scale which ranges from 0 to 6. A score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment. ACQ-IA total score is calculated as the mean of the responses to all 7 questions.
  The measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Weeks 24 and 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a Scale
  Week 24 (N=126, 131, 134) | 1.017 (0.062) | 0.897 (0.060) | 0.835 (0.060)
  Week 48 (N=124, 130, 130) | 0.817 (0.062) | 0.752 (0.060) | 0.723 (0.061)
Statistical Analysis 1: Comparison: Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0975, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.120, 95% CI 2-sided [-0.262 to 0.022], Standard Error of Mean 0.072 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0116, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.182, 95% CI 2-sided [-0.323 to -0.041], Standard Error of Mean 0.072 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.3732, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.065, 95% CI 2-sided [-0.208 to 0.078], Standard Error of Mean 0.073 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.1985, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.093, 95% CI 2-sided [-0.236 to 0.049], Standard Error of Mean 0.073 — Difference calculated as Tio R5 minus placebo

19. Secondary Outcome: ACQ-IA Responder Analysis
Description: Responder categories based on the ACQ-IA total score after 24 and 48 weeks of treatment. Analysis was performed using the following categories and definitions: responder (change from trial baseline ≤-0.5), no change (-0.5 <change from trial baseline <0.5) and worsening (change from trial baseline ≥0.5). No statistical testing was performed for ACQ-IA total score responders.
  The ACQ-IA is a scale containing 7 questions, each question has a 7-point scale which ranges from 0 to 6; a score of 0 corresponds to no impairment and a score of 6 corresponds to maximum impairment.
Time Frame: Weeks 24 and 48
Population: FAS, missing data for patients not withdrawn from the study were either categorised as no change or based on available data, withdrawn patients were imputed based upon discontinuation reason
Measure: Number; unit: Patients
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Patients
  Responders at Week 24 | 97 | 108 | 118
  No Change at Week 24 | 34 | 27 | 16
  Worsening at Week 24 | 0 | 0 | 1
  Responder at Week 48 | 114 | 118 | 117
  No Change at Week 48 | 16 | 14 | 17
  Worsening at Week 48 | 1 | 3 | 1

20. Secondary Outcome: PAQLQ(S) Total Score
Description: Standardised Paediatric Asthma Quality of Life Questionnaire (PAQLQ(S)) total score at weeks 24 and 48.
  The PAQLQ(S) is 23 questions on a 7-point scale, ranging from 1 (worst control) to 7 (best control). Total Score is calculated as mean of all 23 questions.
  The measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Weeks 24 and 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a Scale
  Week 24 (N= 126, 131, 134) | 5.966 (0.065) | 6.142 (0.063) | 6.093 (0.062)
  Week 48 (N=124, 130, 130) | 6.309 (0.065) | 6.288 (0.063) | 6.327 (0.063)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0144, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.176, 95% CI 2-sided [0.035 to 0.316], Standard Error of Mean 0.072 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0747, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.127, 95% CI 2-sided [-0.013 to 0.267], Standard Error of Mean 0.071 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.7654, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.021, 95% CI 2-sided [-0.163 to 0.120], Standard Error of Mean 0.072 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.8082, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.017, 95% CI 2-sided [-0.124 to 0.158], Standard Error of Mean 0.072 — Difference calculated as Tio R5 minus placebo

21. Secondary Outcome: PAQLQ(S) Symptom Domain Score
Description: PAQLQ(S) symptom domain score at weeks 24 and 48. The PAQLQ(S) is 23 questions on a 7-point scale, ranging from 1 (worst control) to 7 (best control). The individual domain score was calculated as the mean of the items in the domain.
  The measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Weeks 24 and 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a Scale
  Week 24 (N=126, 131, 134) | 5.840 (0.076) | 6.015 (0.074) | 5.967 (0.073)
  Week 48 (N=124, 130, 130) | 6.195 (0.076) | 6.177 (0.074) | 6.199 (0.074)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0392, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.175, 95% CI 2-sided [0.009 to 0.341], Standard Error of Mean 0.085 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.1351, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.126, 95% CI 2-sided [-0.039 to 0.292], Standard Error of Mean 0.084 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.8291, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.018, 95% CI 2-sided [-0.185 to 0.149], Standard Error of Mean 0.085 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.9655, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.004, 95% CI 2-sided [-0.163 to 0.171], Standard Error of Mean 0.085 — Difference calculated as Tio R5 minus placebo

22. Secondary Outcome: PAQLQ(S) Activity Limitation Domain Score
Description: PAQLQ(S) activity limitation domain score at weeks 24 and 48. The PAQLQ(S) is 23 questions on a 7-point scale, ranging from 1 (worst control) to 7 (best control). The individual domain score is calculated as the mean of the items in this domain.
  The measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Weeks 24 and 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a Scale
  Week 24 (N= 126, 131, 134) | 5.898 (0.069) | 6.089 (0.067) | 6.023 (0.067)
  Week 48 (N=124, 130, 130) | 6.249 (0.070) | 6.284 (0.068) | 6.319 (0.067)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0139, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.191, 95% CI 2-sided [0.039 to 0.343], Standard Error of Mean 0.077 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.1043, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.125, 95% CI 2-sided [-0.026 to 0.276], Standard Error of Mean 0.077 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.6547, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.035, 95% CI 2-sided [-0.118 to 0.187], Standard Error of Mean 0.078 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.3648, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.070, 95% CI 2-sided [-0.082 to 0.222], Standard Error of Mean 0.077 — Difference calculated as Tio R5 minus placebo

23. Secondary Outcome: PAQLQ(S) Emotional Function Domain Score
Description: PAQLQ(S) emotional function domain score at weeks 24 and 48. The PAQLQ(S) is 23 questions on a 7-point scale, ranging from 1 (worst control) to 7 (best control). The individual domain score is calculated as the mean of the items in this domain.
  The measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Weeks 24 and 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a Scale
  Week 24 (N=126, 131, 134) | 6.157 (0.067) | 6.323 (0.065) | 6.298 (0.064)
  Week 48 (N=124, 130, 130) | 6.481 (0.067) | 6.420 (0.065) | 6.491 (0.065)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.0256, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.166, 95% CI 2-sided [0.020 to 0.312], Standard Error of Mean 0.074 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0561, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.141, 95% CI 2-sided [-0.004 to 0.286], Standard Error of Mean 0.074 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.4127, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.061, 95% CI 2-sided [-0.208 to 0.085], Standard Error of Mean 0.075 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.8922, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.010, 95% CI 2-sided [-0.136 to 0.156], Standard Error of Mean 0.074 — Difference calculated as Tio R5 minus placebo

24. Secondary Outcome: Responders in PAQLQ(S) at Weeks 24 and 48
Description: Responders in PAQLQ(S) at weeks 24 and 48. Analysis was performed using the following categories and definitions: responder (change from trial baseline ≥0.5), no change (-0.5 <change from trial baseline <0.5) and worsening (change from trial baseline ≤-0.5). No statistical testing was performed for PAQLQ(S) total score responders.
  The PAQLQ(S) is 23 questions on a 7-point scale, ranging from 1 (worst control) to 7 (best control).
Time Frame: Weeks 24 and 48.
Population: as for outcome 19
Measure: Number; unit: Patients
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Patients
  Responders at Week 24 | 67 | 82 | 73
  No Change at Week 24 | 58 | 47 | 56
  Worsening at Week 24 | 6 | 6 | 6
  Responders at Week 48 | 89 | 96 | 92
  No Change at Week 48 | 39 | 33 | 42
  Worsening at Week 48 | 3 | 6 | 1

25. Secondary Outcome: Change From Baseline in Nighttime Awakenings
Description: Change from baseline in nighttime awakenings based on the weekly mean at weeks 24 and 48.
  Nighttime awakenings was assessed by the question "Did you wake up during the night due to your asthma?" from the e-diary. Scores range from 1 (did not wake up) to 5 (was awake all night).
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a scale
  Week 24 (N=122, 130, 130) | -0.070 (0.030) | -0.079 (0.029) | -0.144 (0.029)
  Week 48 (N=119, 122, 125) | -0.101 (0.030) | -0.131 (0.029) | -0.127 (0.029)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.7931, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.009, 95% CI 2-sided [-0.080 to 0.061], Standard Error of Mean 0.036 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0369, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.075, 95% CI 2-sided [-0.145 to -0.005], Standard Error of Mean 0.036 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.4086, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.030, 95% CI 2-sided [-0.101 to 0.041], Standard Error of Mean 0.036 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.4714, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.026, 95% CI 2-sided [-0.097 to 0.045], Standard Error of Mean 0.036 — Difference calculated as Tio R5 minus placebo

26. Secondary Outcome: Change From Baseline in Morning Asthma Symptoms
Description: Change from baseline in morning asthma symptoms based on the weekly mean at weeks 24 and 48.
  Morning asthma symptoms was assessed by the question "how were your asthma symptoms this morning?" from the e-diary. Scores range from 1 (no asthma symptoms) to 5 (very severe asthma symptoms).
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a scale
  Week 24 (N=122, 130, 130) | -0.138 (0.039) | -0.138 (0.038) | -0.220 (0.038)
  Week 48 (N=119, 122, 125) | -0.177 (0.039) | -0.230 (0.038) | -0.221 (0.038)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.9880, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.001, 95% CI 2-sided [-0.091 to 0.092], Standard Error of Mean 0.047 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0794, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.082, 95% CI 2-sided [-0.173 to 0.010], Standard Error of Mean 0.046 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.2623, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.053, 95% CI 2-sided [-0.145 to 0.040], Standard Error of Mean 0.047 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.3552, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.043, 95% CI 2-sided [-0.136 to 0.040], Standard Error of Mean 0.047 — Difference calculated as Tio R5 minus placebo

27. Secondary Outcome: Change From Baseline in Daytime Asthma Symptoms
Description: Change from baseline in daytime asthma symptoms based on the weekly mean at weeks 24 and 48.
  Daytime asthma symptoms was assessed by the question "how were your asthma symptoms during the day?" from the e-diary. Scores range from 1 (no asthma symptoms) to 5 (very severe asthma symptoms).
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a scale
  Week 24 (N=121, 130, 133) | -0.204 (0.041) | -0.243 (0.040) | -0.263 (0.040)
  Week 48 (N=119, 123, 125) | -0.261 (0.042) | -0.272 (0.041) | -0.312 (0.041)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.4359, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.039, 95% CI 2-sided [-0.135 to 0.058], Standard Error of Mean 0.049 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.2293, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.059, 95% CI 2-sided [-0.155 to 0.037], Standard Error of Mean 0.049 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.8372, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.010, 95% CI 2-sided [-0.108 to 0.088], Standard Error of Mean 0.050 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.3022, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.051, 95% CI 2-sided [-0.148 to 0.046], Standard Error of Mean 0.049 — Difference calculated as Tio R5 minus placebo

28. Secondary Outcome: Change From Baseline in Daytime Activity Limitations
Description: Change from baseline in daytime activity limitations based on the weekly mean at weeks 24 and 48.
  Daytime activity limitations was assessed by the question "how limited were you in your activities today because of your asthma?" from the e-diary. Scores range from 1 (not limited) to 5 (totally limited).
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a scale
  Week 24 (N=121, 130, 133) | -0.181 (0.039) | -0.212 (0.038) | -0.240 (0.038)
  Week 48 (N=119, 123, 125) | -0.227 (0.039) | -0.238 (0.038) | -0.259 (0.038)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.5004, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.031, 95% CI 2-sided [-0.122 to 0.060], Standard Error of Mean 0.046 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.1982, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.059, 95% CI 2-sided [-0.149 to 0.031], Standard Error of Mean 0.046 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.8019, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.012, 95% CI 2-sided [-0.103 to 0.080], Standard Error of Mean 0.047 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.4872, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.032, 95% CI 2-sided [-0.123 to 0.059], Standard Error of Mean 0.046 — Difference calculated as Tio R5 minus placebo

29. Secondary Outcome: Change From Baseline in Daytime Experiences of Shortness of Breath
Description: Change from baseline in daytime experiences of shortness of breath based on the weekly mean at weeks 24 and 48.
  Daytime experiences of shortness of breath was assessed by the question "how much shortness of breath did you experience during the day" from the e-diary. Scores range from 1 (none) to 5 (a very great deal).
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a scale
  Week 24 (N=121, 130, 133) | -0.134 (0.039) | -0.178 (0.038) | -0.240 (0.038)
  Week 48 (N=119, 123, 125) | -0.219 (0.039) | -0.231 (0.038) | -0.253 (0.038)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.3498, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.043, 95% CI 2-sided [-0.135 to 0.048], Standard Error of Mean 0.046 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0222, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.106, 95% CI 2-sided [-0.196 to -0.015], Standard Error of Mean 0.046 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.7990, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.012, 95% CI 2-sided [-0.104 to 0.080], Standard Error of Mean 0.047 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.4586, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.035, 95% CI 2-sided [-0.126 to 0.057], Standard Error of Mean 0.047 — Difference calculated as Tio R5 minus placebo

30. Secondary Outcome: Change From Baseline in Daytime Experiences of Wheeze or Cough
Description: Change from baseline in daytime experiences of wheeze or cough based on the weekly mean at weeks 24 and 48.
  Daytime experiences of wheeze or cough was assessed by the question "did you experience wheeze or cough during the day?" from the e-diary. Scores range from 1 (not at all) to 5 (all the time).
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Units on a scale
  Week 24 (N=121, 130, 133) | -0.261 (0.046) | -0.307 (0.045) | -0.355 (0.045)
  Week 48 (N=119, 123, 125) | -0.340 (0.047) | -0.337 (0.045) | -0.393 (0.046)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.4221, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.045, 95% CI 2-sided [-0.156 to 0.065], Standard Error of Mean 0.056 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.0959, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = -0.093, 95% CI 2-sided [-0.204 to 0.017], Standard Error of Mean 0.056 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.9627, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.003, 95% CI 2-sided [-0.109 to 0.114], Standard Error of Mean 0.057 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.3457, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = -0.054, 95% CI 2-sided [-0.165 to 0.058], Standard Error of Mean 0.057 — Difference calculated as Tio R5 minus placebo

31. Secondary Outcome: Change From Baseline in Asthma Symptom-free Days
Description: Change from baseline in asthma symptom-free days based on the weekly mean at weeks 24 and 48.
  A day was considered as an asthma symptom-free day if there were no symptoms reported via the e-Diary (electronic diary) and no use of rescue medication reported via the eDiary during that day.
  Measured values presented are actually adjusted means.
  The number of participants analysed displays the number of participants included in the statistical model whereas the N's for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline and Week 24, Baseline and Week 48.
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Days
Arm/Group | Placebo Respimat | Tio R2.5 | Tio R5
Number analyzed (Participants) | 131 | 135 | 135
Days
  Week 24 (N=122, 130, 133) | 0.135 (0.036) | 0.176 (0.034) | 0.172 (0.035)
  Week 48 (N=120, 123, 127) | 0.151 (0.036) | 0.170 (0.035) | 0.180 (0.035)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tio R2.5; Week 24; Test type: Superiority or Other; p = 0.3375, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.041, 95% CI 2-sided [-0.043 to 0.125], Standard Error of Mean 0.043 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 2: Comparison: Placebo Respimat vs Tio R5; Week 24; Test type: Superiority or Other; p = 0.3880, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Mean Difference (Net) = 0.037, 95% CI 2-sided [-0.047 to 0.121], Standard Error of Mean 0.043 — Difference calculated as Tio R5 minus placebo
Statistical Analysis 3: Comparison: Placebo Respimat vs Tio R2.5; Week 48; Test type: Superiority or Other; p = 0.6541, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.019, 95% CI 2-sided [-0.066 to 0.104], Standard Error of Mean 0.043 — Difference calculated as Tio R2.5 minus placebo
Statistical Analysis 4: Comparison: Placebo Respimat vs Tio R5; Week 48; Test type: Superiority or Other; p = 0.5089, Mixed Models Analysis; Repeated measures restricted maximum likelihood model; Median Difference (Net) = 0.028, 95% CI 2-sided [-0.056 to 0.133], Standard Error of Mean 0.043 — Difference calculated as Tio R5 minus placebo

ADVERSE EVENTS:
Time Frame: From first drug intake until 30 days after last drug intake, up to day 407.
Groups:
- Placebo: Inhalation of placebo solution (2 puffs) once daily for 48 weeks delivered by the Respimat inhaler, as add on therapy on top of usual care.
Arm/Group | Placebo | Tio R2.5 | Tio R5
Serious Adverse Events (participants affected / at risk) | 6/131 | 3/135 | 1/135
Other Adverse Events (participants affected / at risk) | 79/131 | 76/135 | 71/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=131) | Tio R2.5 (N=135) | Tio R5 (N=135)
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Renal abscess (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Paranasal sinus haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=131) | Tio R2.5 (N=135) | Tio R5 (N=135)
Nasopharyngitis (Infections and infestations) | 13 | 15 | 12
Rhinitis (Infections and infestations) | 7 | 5 | 2
Peak expiratory flow rate decreased (Investigations) | 27 | 31 | 29
Asthma (Respiratory, thoracic and mediastinal disorders) | 57 | 49 | 46
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 6
Respiratory tract infection (Infections and infestations) | 16 | 11 | 13
Respiratory tract infection viral (Infections and infestations) | 8 | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.